CLINICAL TRIAL: NCT07341412
Title: Clinical and Genetic Aspects in Fetuses and Children With Sex Chromosome Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-65-24
Record Dates: First submitted 2025-12-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Sex Chromosome Disorders
Keywords: Turner syndrome; Klinefelter syndrome; Triple X syndrome; Double Y syndrome; 45,X/46,XY syndrome
MeSH Terms: conditions — Sex Chromosome Disorders; Turner Syndrome; Klinefelter Syndrome; Triple X syndrome; XYY Karyotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, saliva, urine, feces, placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Pregnant women carrying a fetus with a sex chromosome disorder
- Pregnant women carrying a fetus without a sex chromosome disorder (Controls)
- Mothers of a child with a sex chromosome disorder
- MOthers of a child without a sex chromosome disorder (Controls)
- Children with a sex chromosome disorder
- Children without a sex chromosome disorder (Controls)

SUMMARY:
The aim of the project is to:

1. Investigate organ development and growth in fetuses with sex chromosome disorders;
2. Investigate growth, development, and morbidity in children with sex chromosome disorders during the first years of life;
3. Delineate how variations in sex chromosome number affect the epigenetic and genetic mechanisms regulating gene expression in the placenta and in multiple tissues of the child after birth over time during early childhood;
4. Investigate the gut microbiome in children with sex chromosome disorders during the first years of life;
5. Identify the epigenetic and genetic mechanisms and placental and child-specific alterations underlying the phenotype observed in fetuses, children, and adults with sex chromosome disorders, using a deep phenotyping approach.

ELIGIBILITY:
Inclusion Criteria for pregnant participants in case group:

Age ≥18 years Fetus with a genetically verified sex chromosome disorder Written informed consent

Inclusion Criteria for pregnant participants in control group:

Age ≥18 years Normal first- and second-trimester ultrasound examinations Fetal growth within the normal range Written informed consent

Inclusion Criteria for mothers in the case group:

Age ≥18 years at the time of pregnancy with the child Child with a genetically verified sex chromosome disorder Written informed consent

Inclusion Criteria for mothers in the control group:

Age ≥18 years at the time of pregnancy with the child Normal first- and second-trimester ultrasound examinations during the pregnancy Normal fetal growth during the pregnancy Written informed consent

Inclusion Criteria for children in the case group:

If parents share joint custody, written informed consent must be obtained from both parents Ability to undergo a physical examination Child with a genetically verified sex chromosome disorder (prenatally or postnatally diagnosed)

Inclusion Criteria for children in the control group:

If parents share joint custody, written informed consent must be obtained from both parents Ability to undergo a physical examination

Exclusion Criteria for all groups:

Severe claustrophobia Implanted magnetic material contraindicating MRI

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Recruitment of cases will take place at obstetric departments, departments of clinical genetics, and pediatric departments throughout Denmark.
  Recruitment of controls will take place at the Department of Gynecology and Obstetrics and Department of Pediatrics, Aarhus University Hospital as well as via Facebook groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Level of DNA methylation | 5 years
  Levels of DNA methylation in placenta, blood, saliva, and urothelial cells
Level of RNA ekspression | 5 years
  Level of RNA ekspression in placenta, blood, saliva, and urothelial cells
Height | 5 years
  Height in centimeter (cm)
Weight | 5 years
  Weight in kilogram (kg) or gram (g)
Body mass index | 5 years
  Body mass index (BMI) in kg/m²
Head circumference | 5 years
  head circumference in centimeter (cm)
Fat mass and fat-free mass | 5 years
  Measure of fat mass and fat-free mass by PEA POD (kg)
Development | 5 years
  Bayley-4 will be used to measure development. Ages & Stages Questionnaires will be used to measure development including social-emotional development drawing on the parents knowledge.
Fecal microbial diversity | 5 years
  Measure of fecal microbial diversity
Fecal microbial composition | 5 year
  Measurement of fecal microbial composition
Left ventricular ejection fraction | 5 years
  Left ventricular ejection fraction measured by echocardiography (%)
Left ventricular diameters | 5 years
  Left ventricular end-diastolic and end-systolic diameters measured by echocardiography (mm)
Interventricular septal wall thickness | 5 years
  Interventricular septal wall thickness measured by echocardiography (mm)
Heart rate | 5 years
  Heart rate (beats per minute) measured by electrocardiogram
PR interval | 5 years
  PR interval (ms) measured by electrocardiogram
QRS duration | 5 years
  QRS duration (ms) measured by electrocardiogram
Corrected QT interval | 5 years
  Corrected QT interval (ms) measured by electrocardiogram
Blood pressure | 5 years
  Systolic and diastolic blood pressure (mmHg)
Congenital heart malformation | 5 years
  Congenital heart malformation assessed by echocardiography
Aorta diameter | 5 years
  Aorta diameter (mm) measured by echocardiography
Aortic valve mean gradient | 5 years
  Measure of aortic valve mean gradient (mmHG)
Mitral valve mean gradient | 5 years
  Measure of mitral valve mean gradient (mmHg)
Transaortic doppler flow | 5 years
  Measure of transaortic doppler flow (m/s)
Fetal brain volume | 5 years
  Fetal brain volume measured by MRI (cm³)
Fetal heart volume | 5 years
  Fetal heart volume measured by MRI (cm³)
Fetal kidney volume | 5 years
  Fetal kidney volume measured by MRI (cm³)
Fetal lever volume | 5 years
  Fetal lever volume measured by MRI (cm³)
Fetal spleen volume | 5 years
  Fetal spleen volume measured by MRI (cm³)
Fetal gonadal volume | 5 years
  Fetal gonadal volume measured by MRI (cm³)

SECONDARY OUTCOMES:
Left ventricular mass | 5 years
  Calculation of left ventricular mass (g)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Skakkebæk, MD, PHD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No